CLINICAL TRIAL: NCT03547596
Title: Impact of Treatment of Obstructive Sleep Apnea Syndrome by Continuous Positive Airway Pressure Equipment at Night on the Lower Urinary Tract Symptoms and the Erectile Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO18063
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-05

CONDITIONS: Lower Urinary Tract Symptoms; Erectile Dysfunction; Obstructive Sleep Apneas Syndrom
Keywords: Lower urinary tract symptoms; Erectile dysfunction; Obstructive Sleep Apneas Syndrom
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire passation — Questionnaires to evaluate lower urinary tract symptoms and erectile dysfunction.

SUMMARY:
To treat lower urinary tract symptoms (LUTS) and erectile dysfunction (ED), we mainly have symptomatic drug treatments. Some patients are resistant to the treatments that we have or are forced to stop treatments because of side effects.

It would be interesting to focus on comorbidities and to evaluate whether it is possible to improve the urological symptoms by taking care the comorbidities, which would consist in an etiological treatment of the urological symptoms.

The aim of the study is to evaluate the evolution of low urinary tract disorders (LUTS) and erectile dysfunction (ED) in patients with obstructive sleep apnea syndrome (OSAS) following by continuous positive airway pressure equipment (CPAP) at night.

Participation in the study will be offered to all patients, men and women, consulting or hospitalized in the sleep unit of the department of pneumology CHU of Reims for a nocturnal ventilatory polygraphy or a polysomnography diagnostic of OSAS.

Men will complete three questionnaires about LUTS and DE, women one questionnaire about LUTS. The questionnaires will be completed twice, the first time when consulting at the sleep unit for nocturnal ventilatory polygraphy or a polysomnography diagnostic of OSAS ; the second time during the pneumology consultation three months later. We will compare the results between the questionnaires to assess whether OSAS equipment with CPAP has improved urologic symptoms.

If the management of OSAS allows an improvement of lower urinary tract disorders and / or an improvement of erectile dysfunction, these results would be interesting for the management of patients resistant to symptomatic drug treatments or to stop them because of iatrogenic side effects.

Etiological rather than symptomatic management would also have long-term benefits, both in improving the overall quality of life of the patient and in the medical and economic field.

It might be interesting to identify in urology consultation among patients consulting for LUTS or ED, patients at risk of presenting OSAS and referring them to a pulmonologist to manage OSAS if it exists, from the beginning of the urological care.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is the most common nocturnal breathing disorder. It is characterized by the occurrence, during sleep, of repeated episodes of complete collapse (apnea) or incomplete (hypopneas) of the upper airways. OSAS is a pathology that, through its cardiovascular and metabolic complications, its impact on daytime vigilance, represents a real public health problem. The prevalence of OSA is estimated at 2% in women and 4% in men aged 30 to 60 years. Recent studies estimate that nearly 2 million French people will be affected by this pathology.

The lower urinary tract symptoms (LUTS) include: disorders of the filling phase (urinary incontinence, diurnal and nocturnal pollakiuria, nocturia, urgency), disorders of the urinary phase, dysuria (weakness of the jet, urination by pushing, urinary burns), symptoms of the post-mictionnal phase (incomplete bladder emptying sensation).

LUTS have several etiologies. Dysuria is cause by obstacle under vesical (benign prostatic hyperplasia, urethral stenosis, bladder neck disease), neurological bladder, genital prolapse, drug etiology (parasympatholytic). Concerning pollakiuria and urgency there are bladder etiologies (cystitis, foreign body, tumor, neurological bladder), sub-bladder obstruction, extra-vesical etiologies (infectious pathology of contact, pregnancy, extrinsic tumor compression).

LUTS are responsible for an alteration of the quality of life. In men, LUTS are often caused by benign prostatic hypertrophy (BPH), which is one of the most common conditions in men over 40 years of age. The prevalence of BPH is variable in the literature: in men over 50 years of age with moderate symptomatology, the prevalence is of the order of 25%, it is estimated at 50 to 75% for men 65 years and over.

The prevalence of overactive bladder is estimated at 14.4% in France, it increases with age and among women.

Erectile dysfunction (ED) is the inability to obtain and / or maintain an erection sufficient to allow satisfactory sexual activity; for at least 3 months.

The prevalence of ED is high, it affects one in three men after the age of 40 and has a significant impact on the quality of life of patients. The appearance of an ED must make search for cardiovascular diseases. The prevalence of ED increases with co-morbidities such as high blood pressure, diabetes, dyslipidemia, obesity and smoking.

To treat lower urinary tract symptoms (LUTS) and erectile dysfunction (ED), we mainly have symptomatic drug treatments. Some patients are resistant to the treatments that we have or are forced to stop treatments because of side effects. It would be interesting to focus on comorbidities and to evaluate whether it is possible to improve the urological symptoms by taking care the comorbidities, which would consist in an etiological treatment of the urological symptoms.

The aim of the study is to evaluate the evolution of low urinary tract disorders (LUTS) and erectile dysfunction (ED) in patients with obstructive sleep apnea syndrome (OSAS) following by continuous positive airway pressure equipment (CPAP) at night.

Participation in the study will be offered to all patients, men and women, consulting or hospitalized in the sleep unit of the department of pneumatology CHU Reims for nocturnal ventilation polygraphy or diagnostic polysomnography of OSAS.

Information about the purpose and modalities of the study will be given to the patient by a pulmonologist or urologist using an information note. If the patient agrees to participate in the study (signing the non-objection form), he / she will be included in the study.

Participation in the study will consist of:

* a filling of questionnaires on LUTS : Urinary Symptom Profil (USP) for all patients, International Prostate Score Symptoms (IPSS) only for men and disorders of erectile function International Index of Erectile Function (IIEF5) for men during hospitalization for a nocturnal ventilatory polygraphy or a diagnostic polysomnography of OSAS.

The criterion for polysomnography is the hypopnoea apnea index (HAI) which is defined as the number of apneas and hypopneas per hour. The diagnosis of OSAS is confirmed if, in addition to the clinical symptoms, the HAI is >5 events per hour. The severity of OSAS is defined according to the HAI: the OSAS is moderate if the HAI is >15 events per hour, the OSAS is severe if HAI >30 events per hour.

IPSS, USP and IIEF5 are international questionnaires, recognized and validated by the French Association of Urology.

The IPPS questionnaire is only for men and has 7 items on lower urinary tract disorders and an item on quality of life. Each item is rated between 0 and 5 depending on the frequency of the disorders. The score is the sum of the items. The symptoms are mild if the score is between 0 and 7, moderate if the score is between 8 and 19, severe if the score is between 20 and 35.

The USP questionnaire is validated psychometrically. It is intended for men and women.

It includes an item on stress urinary incontinence, 6 items on bladder hyperactivity and 3 items on dysuria. Each item is scored between 0 and 3 depending on the severity of the symptoms. The score for each symptom is the sum of the corresponding items.

The IIEF5 questionnaire is intended for men only. It has 5 items on erectile dysfunction.

Each item is rated between 0 and 5 depending on the severity of the symptoms. Erectile function is normal if the score is between 21 and 25.The erectile dysfunction is mild if the score is between 16 and 20, moderate if the score is between 11 and 15, severe if the score is between 5 and 10, and not interpretable if the score is between 0 and 4.

* a collection of data concerning the patient (sex, age, tobacco), his comorbidities (weight, height and body mass index, hypertension, diabetes, hypercholesterolemia, myocardial infarction, stroke, anxiety and / or depression) and his treatment (including drug classes that may interact with urologic symptoms: antihypertensives, diuretics, alpha blockers, 5 alpha-reductase inhibitors, phosphodiesterase type 5 inhibitors, herbal medicine).

In addition, patients with moderate or severe OSAS (not warranting implementation of nocturnal CPAP therapy) as well as moderate or severe urological symptoms objected to by the questionnaires (IPSS> 7 and / or USP not 0 + 0 + 0 and / or IIEF5 ≤ 20) will again complete the questionnaires on lower urinary tract disorders and disorders of erectile function during the follow-up consultation in pulmonology post PPC equipment (at 3 months post equipment or at 6 months post equipment if the observance or the effectiveness of the apparatus is not optimal with M3).

Participation in the study does not change the patient's medical management regarding OSAS.

The duration of participation will be punctual for patients with no moderate or severe OSA associated with moderate or severe urological symptoms. The duration of patient participation will be from 3 months to 6 months for patients with moderate or severe OSAS associated with moderate or severe urological symptoms. This duration of participation corresponds to the time necessary to obtain an observance and an optimal efficiency of the apparatus by PPC allowing to consider a clinical improvement of the disturbances of the sleep.

ELIGIBILITY:
Inclusion criteria :

* managed at the sleep unit at Reims University Hospital for the diagnosis of sleep apnea syndrome by nocturnal airway polygraphy or polysomnography
* major
* accepting participation in the study (signed non-opposition form)

Exclusion criteria :

* refusing to be included in the study
* minors
* not speaking French or not able to read (inability to complete the questionnaires specific to the study).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years, men and women, managed in the sleep unit of Reims University Hospital for the realization of a nocturnal ventilatory polygraphy or polysomnography in search of an OSAS during the inclusion phase and accepting to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-04-29 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
lower urinary tract symptoms | Day 0
  Evaluation of the lower urinary tract symptoms using "UrinarySymptom Profil"
erectile dysfunction | Day 0
  Evaluation of the lower urinary tract symptoms using "International Index of Erectile Function"

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France